CLINICAL TRIAL: NCT07025681
Title: Randomized, Double-blinded, Two-treatment, Two-periods, Single-dose, Crossover, PK, PD, Safety, and Immunogenicity Study of Erythropoietin of Incepta Pharmaceuticals Ltd With Eprex of Janssen-Cilag Ltd in Healthy Adult Subjects
Brief Title: PK, PD, Safety and Immunogenicity Study of Erythropoietin of Incepta Pharmaceuticals Ltd With Eprex (Janssen-Cilag).
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incepta Pharmaceuticals Ltd (Industry)
Collaborators: Institute for Developing Science and Health Initiatives, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/CT/01
Record Dates: First submitted 2025-05-24; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Erythropoietin; cross over; Eprex; Double blinded

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythropoietin 4000 IU Injection of Incepta Pharmaceuticals Ltd (Experimental): Erythropoietin 4000 IU Injection, subcutaneous injection manufactured by Incepta Pharmaceuticals Ltd will be administered.
  Interventions: Biological: Erythropoietin alfa
- Eprex 4000 by Janssen-Cilag Ltd (Active Comparator): Eprex 4000, subcutaneous injection manufactured by Janssen-Cilag Ltd will be administered.
  Interventions: Biological: Erythropoietin alfa

INTERVENTIONS:
Biological: Erythropoietin alfa — Erythropoietin 4000 IU Injection, for subcutaneous injection.

SUMMARY:
Erythropoietin is a glycoprotein which stimulates red blood cell production. It is produced in the kidney and stimulates the division and differentiation of committed erythroid progenitors in the bone marrow. Erythropoietin, a 165 amino acid glycoprotein manufactured by recombinant DNA technology, has the same biological effects as endogenous erythropoietin. Erythropoietin binds to the surface receptor of erythroid precursor cells and activates signal transduction pathways that interfere with apoptosis and stimulates erythroid cell proliferation. Recombinant human erythropoietin is a substitute for the deficiency observed in CKD, therapy of anemia often involves many other issues such as Anemia in patients with non-myeloid malignancies where anemia is due to the effect of concomitantly administered chemotherapy, Anemic patients (hemoglobin > 10 to < 13 g/dL) scheduled to undergo elective, noncardiac, nonvascular surgery to reduce the need for allogeneic blood transfusions, Anemia related to therapy with zidovudine in HIV-infected patients are also needed to be considered in order to effectively correct anemia, reduce costs and minimize side effects.

DETAILED DESCRIPTION:
In this study, 56 healthy adult volunteers will participate in a randomized, double-blinded, balanced, two-treatment, two-period, two-sequence, single-dose crossover trial. Each subject will receive a single subcutaneous injection of either Erythropoietin 4000 IU manufactured by Incepta Pharmaceuticals Ltd (test product) or Eprex 4000 IU manufactured by Janssen-Cilag Ltd (reference product) under fasting conditions, with a 28-day washout period between doses. The primary aim of the study is to compare the pharmacokinetic and pharmacodynamic profiles of the two products. Additionally, the study will assess immunogenicity by measuring serum anti-drug antibodies (ADA) and evaluate the safety of both formulations throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years.

  * BMI of 18.0-30.0kg/m2.
  * Voluntarily participants who agree to observe the precautions in writing after receiving a complete explanation of this trial.
  * Willingness and ability to undertake all scheduled visits and assessments.
  * Subject who have no evidence of underlying disease during screening, medical history and whose physical examination is performed within 28 days prior to commencement of the study.
  * Subjects whose screening laboratory values are within normal limits or considered by the Investigator to be of no clinical significance.
  * Non-smokers, ex-smokers and light smokers can be included in the study. "Light smokers are defined as someone smoking < 10 cigarettes per day, ex-smokers as someone who completely stopped smoking for at least 03 months.
  * No alcohol dependence, alcohol abuse or drug abuse (Amphetamines, Cocaine, Tetra Hydro Cannabinoids, Benzodiazepines, Barbiturates and Opioids) within the past one year.
  * Subjects should not have consumed grape fruit juice or its products 72 hours before dosing and throughout the study periods.
  * For Female Subjects:

    1. Subjects having negative urine pregnancy test.
    2. Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the Investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
    3. Postmenopausal for more than 1 year.
    4. Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

* • Subjects with any previous exposure to erythropoiesis stimulating agents.

  * History of clinically significant illness related to liver (including viral hepatitis), kidney, nervous system, immune system, respiratory system, endocrine system, cardiovascular system, blood system and tumor as well as mental illness (mood disorder, obsessive-compulsive disorder, etc.)
  * Hypersensitivity or clinically significant hypersensitivity to the drug (e.g. aspirin, antibiotics, etc.)
  * Those whose results meet more than one of the followings in the screening including re-test; Hemoglobin level below 12g/dL or over 17g/dL, Ferritin level below 21.8ng/mL, Transferrin level below 190mg/dL, Reticulocyte level >2.5%, erythrocytes level > 5.2x 106/mm3, platelets or serum potassium level over normal range.
  * Positive on the HIV antibody, HBsAg, HCV (Hepatitis C Virus) antibody tests.
  * Those whose vital signs measured in sitting position after resting over 3 minutes meet more than one of the following; Systolic BP below 90mmHg or over 160mmHg, Diastolic BP below 50mmHg or over 100mmHg, Pulse rate over 100.
  * Those who received the following diagnosis within 6 months prior to the screening; Hemoglobinopathy (e.g., homozygous sickle-cell disease, thalassemia of all kinds), Chronic or uncontrollable inflammatory diseases (e.g., rheumatoid arthritis, systemic erythematosus)
  * Those who participated other clinical trials and was administered other drugs within 3 months prior to the scheduled dose.
  * Those who bled over 400mL or donated blood within 8 weeks prior to the scheduled first dose.
  * Those who are considered inappropriate for the trial by the trial investigator based on the result of clinical laboratory test or due to other reasons.
  * Employees of Investigational sites, individuals directly involved with the conduct of the study or immediate family members thereof, prisoners, and persons who are legally institutionalized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 144.00±1* hours following drug administration after each dose.
  The PK parameter Cmax shall be calculated by noncompartmental analysis using Phoenix® WinNonlin. The maximum observed serum EPO concentration (Cmax) shall be directly obtained from the data.
Reticulocyte count (%) | 312±1 hours post dose.
  As primary PD parameter, maximum effect change (Delta Emax) and the area under the baseline-adjusted effect curve (Delta AUEC) shall be calculated by the linear trapezoidal method for the RET count.
Area under the plasma concentration versus time curve (AUC) | 144.00±1* hours following drug administration
  The PK parameters shall be calculated by noncompartmental analysis using Phoenix® WinNonlin. The maximum observed serum EPO concentration (Cmax) and the time of Cmax (Tmax) shall be directly obtained from the data. The AUClast shall be calculated by the linear trapezoidal method up to Tmax and by the log trapezoidal method after Tmax. The area under the curve extrapolated to infinity (AUCinf) shall be obtained with the following formula: AUCinf=AUClast+Clast, where Clast is the last observed serum EPO concentration and lambda z is a calculated terminal elimination rate constant.

SECONDARY OUTCOMES:
t1/2 | 144.00±1* hours following drug administration.
  The terminal half-life (t1/2) shall be calculated by dividing natural-log2 by lambda z.
Immunogenicity | At 00.00 hours of period I and at 312±1 hours post dose of period II
  By measuring Anti-drug Antibody (ADA) formation.
Hemoglobin | From baseline and up to 312±1 hours following drug administration
  Mean absolute change in Hb levels between the baseline period (pre dose) and the evaluation period.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Umme Kulsum, Principal Investigator — Institute for developing Science and Health initiatives (ideSHi), Dhaka-1206, Bangladesh
Locations (1):
- Universal Medical College and Hospital, Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
By publication in the journal
Supporting Information: Study Protocol, CSR
Time Frame: After completion of study
Access Criteria: Journal

REFERENCES:
- [Background] Yan X, Lowe PJ, Fink M, Berghout A, Balser S, Krzyzanski W. Population pharmacokinetic and pharmacodynamic model-based comparability assessment of a recombinant human Epoetin Alfa and the Biosimilar HX575. J Clin Pharmacol. 2012 Nov;52(11):1624-44. doi: 10.1177/0091270011421911. Epub 2011 Dec 12. PMID 22162538
- [Background] Yoon S, Rhee SJ, Heo SJ, Oh TY, Yoon SH, Cho JY, Lee S, Yu KS. Comparable pharmacokinetics and pharmacodynamics of two epoetin alfa formulations Eporon(R) and Eprex(R) following a single subcutaneous administration in healthy male volunteers. Drug Des Devel Ther. 2017 Oct 27;11:3127-3135. doi: 10.2147/DDDT.S142673. eCollection 2017. PMID 29138535
- [Background] Elliott S, Pham E, Macdougall IC. Erythropoietins: a common mechanism of action. Exp Hematol. 2008 Dec;36(12):1573-84. doi: 10.1016/j.exphem.2008.08.003. Epub 2008 Oct 14. PMID 18922615
- [Background] Rashidi A, Garimella PS, Al-Asaad A, Kharadjian T, Torres MN, Thakkar J. Anemia Management in the Cancer Patient With CKD and End-Stage Kidney Disease. Adv Chronic Kidney Dis. 2022 Mar;29(2):180-187.e1. doi: 10.1053/j.ackd.2022.03.005. PMID 35817525
- [Background] Portoles J, Martin L, Broseta JJ, Cases A. Anemia in Chronic Kidney Disease: From Pathophysiology and Current Treatments, to Future Agents. Front Med (Lausanne). 2021 Mar 26;8:642296. doi: 10.3389/fmed.2021.642296. eCollection 2021. PMID 33842503
- [Background] Jelkmann W. Physiology and pharmacology of erythropoietin. Transfus Med Hemother. 2013 Oct;40(5):302-9. doi: 10.1159/000356193. Epub 2013 Jul 19. PMID 24273483